CLINICAL TRIAL: NCT07373847
Title: A Single-center, Randomized, Placebo-controlled Trial Study to Compare Efficacy, Safety and Tolerability of Vunakizumab Combined With Recaticimab in Subjects With Moderate to Severe Plaque Psoriasis and Dyslipidemia
Brief Title: Vunakizumab Combined With Recaticimab in Subjects With Moderate to Severe Plaque Psoriasis and Dyslipidemia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA-DER-IV-015
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: adults with moderate-to-severe psoriasis treated by vunakizumab and recaticimab. (Experimental): The recommended dosage of vunakizumab is 240 mg (administered as two 120 mg injections), given subcutaneously at Weeks 0, 2, and 4, followed by maintenance dosing every 4 weeks. For recaticimab, the recommended dosages are 150 mg subcutaneously every 4 weeks or 300 mg every 8 weeks.
  Interventions: Drug: vunakizumab and recaticimab.
- Active Comparator: adults with moderate-to-severe psoriasis treated by vunakizumab and placebo. (Placebo Comparator): The recommended dosage of vunakizumab is 240 mg (administered as two 120 mg injections), given subcutaneously at Weeks 0, 2, and 4, followed by maintenance dosing every 4 weeks. For placebo, the recommended dosages are 150 mg subcutaneously every 4 weeks or 300 mg every 8 weeks.
  Interventions: Drug: vunakizumab and placebo

INTERVENTIONS:
Drug: vunakizumab and recaticimab. — Adult patients (>18 years) with moderate-to-severe psoriasis who will start treatment with either vunakizumab and recaticimab.
  Arms: Active Comparator: adults with moderate-to-severe psoriasis treated by vunakizumab and recaticimab.
Drug: vunakizumab and placebo — Adult patients (>18 years) with moderate-to-severe psoriasis who will start treatment with either vunakizumab and placebo.
  Arms: Active Comparator: adults with moderate-to-severe psoriasis treated by vunakizumab and placebo.

SUMMARY:
The aim is to evaluate the safety and efficacy of vunakizumab combined with recaticimab versus vunakizumab combined with placebo in the treatment of plaque psoriasis with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects who meet all of the following criteria may be enrolled in this study:

Adults aged 18 to 75 years, inclusive.

Clinically confirmed diagnosis of psoriasis.

At screening or on Day 1 of study treatment, a PASI score ≥10, BSA involvement ≥10%, and PGA score ≥3.

Presence of dyslipidemia at screening or on Day 1 of study treatment, defined as fasting LDL-C ≥2.6 mmol/L and <4.9 mmol/L in subjects without concomitant atherosclerotic cardiovascular disease (ASCVD).

Fasting triglycerides (TG) <5.6 mmol/L and 10-year ASCVD risk score <10%.

Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline, and must agree to use effective contraception throughout the study and for 30 days after the end of the study.

Subjects must voluntarily participate in the study and provide written informed consent.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

Presence of non-plaque psoriasis at screening or on Day 1 of the study, including guttate, inverse, pustular, erythrodermic, or drug-induced psoriasis.

Fever or active infection within 7 days prior to study initiation.

History of serious infection within 60 days prior to study initiation (including but not limited to bacterial, viral, or fungal infections requiring hospitalization or intravenous antimicrobial therapy), or any untreated infection.

History of chronic infection, such as chronic pyelonephritis or chronic osteomyelitis.

Positive hepatitis B virus (HBV) DNA with abnormal liver function, or HBV DNA >1 × 10⁵ copies/mL, indicating active infection.

Positive test results for human immunodeficiency virus (HIV) or Treponema pallidum (syphilis) antibodies.

Clinical signs or symptoms suggestive of active tuberculosis (TB) during screening (e.g., fever, cough, night sweats, weight loss), or evidence of current or active pulmonary TB on chest imaging (X-ray or CT) during screening or within 6 months prior to screening.

New York Heart Association (NYHA) class III or IV heart failure, or left ventricular ejection fraction <30%.

Diagnosis within 3 months prior to randomization of new-onset myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass grafting, or stroke.

Type 1 diabetes mellitus, poorly controlled type 2 diabetes mellitus (HbA1c ≥10%), or diabetes with multiple organ comorbidities.

SCORE (Systematic Coronary Risk Evaluation) ≥10%.

During screening, uncontrolled hypertension (defined as systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) or moderate to severe renal impairment, defined as estimated glomerular filtration rate <30 mL/min/1.73 m².

Ongoing active liver disease or liver function abnormalities, defined as ALT and/or AST ≥3× the upper limit of normal (ULN).

Presence of malignancy.

History of severe drug allergy, or known hypersensitivity to funakinzumab, ricazinumab, or any of their excipients.

Pregnant or breastfeeding women, women planning pregnancy during the study period, or male or female subjects unwilling to use contraception.

Receipt of systemic oral or intravenous treatment prior to screening without completion of the required washout period, as defined below:

1. Use of TNF-α, IL-12/23, IL-17, or IL-23 monoclonal antibodies (e.g., adalimumab, ustekinumab, ixekizumab, secukinumab, guselkumab) within 3 months prior to screening;
2. Use of systemic psoriasis treatments (including but not limited to methotrexate, JAK inhibitors, acitretin, cyclosporine, oral or injectable corticosteroids) within 4 weeks prior to screening;
3. Use of topical psoriasis treatments (including but not limited to corticosteroids, vitamin D₃ analogues, calcineurin inhibitors, tapinarof) within 2 weeks prior to screening;
4. Receipt of phototherapy (including oral or topical PUVA, UVB, tanning beds, or therapeutic sun exposure) within 4 weeks prior to screening;
5. Use of statins, cholesterol absorption inhibitors, or fibrates within 4 weeks prior to screening.

Laboratory abnormalities at screening meeting any of the following criteria:

1. Absolute white blood cell count <3,000/mm³;
2. Absolute lymphocyte count <500/mm³;
3. Absolute neutrophil count <1,000/mm³;
4. Platelet count <100,000/mm³;
5. Hemoglobin <9 g/dL;
6. ALT and/or AST >3× ULN;
7. Total unconjugated and/or conjugated bilirubin >2× ULN;
8. Clinically significant electrocardiogram (ECG) abnormalities;
9. Any other laboratory abnormality deemed by the investigator to interfere with study completion or interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
PASI 100 response rate at week 16 in the group treated with vunakizumab combined with recaticimab versus vunakizumab combined with placebo | From enrollment to the end of treatment at 16 weeks

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Yan K, Li F, Bi X, Han L, Zhang Z, Chen R, Li Y, Zhang L, Wang X, Li L, Lu J, Xu A, Yang S, Lu Y, Sun J, Li Z, Zhu X, Jiang M, Zhang S, Wang W, Li Y, Meng Z, Li H, Mou K, Han X, Li S, Chen A, Li X, Liu D, Zhang C, Ji C, Wang Y, Cheng H, Cui X, Yao X, Bai X, Dong G, Xu J. Efficacy and safety of vunakizumab in moderate-to-severe chronic plaque psoriasis: A randomized, double-blind, placebo-controlled phase 3 trial. J Am Acad Dermatol. 2025 Jan;92(1):92-99. doi: 10.1016/j.jaad.2024.09.031. Epub 2024 Sep 26. PMID 39332633
- [Result] Zimerman A, Kunzler ALF, Weber BN, Ran X, Murphy SA, Wang H, Honarpour N, Keech AC, Sever PS, Sabatine MS, Giugliano RP. Intensive Lowering of LDL Cholesterol Levels With Evolocumab in Autoimmune or Inflammatory Diseases: An Analysis of the FOURIER Trial. Circulation. 2025 May 20;151(20):1467-1476. doi: 10.1161/CIRCULATIONAHA.124.072756. Epub 2025 Apr 21. PMID 40255182